CLINICAL TRIAL: NCT03463486
Title: Outpatient Cardiac Rehabilitation in Austria
Brief Title: Current Outpatient Cardiac Rehabilitation in Austria
Status: Completed | Type: Observational
Sponsor: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Prof. Josef Niebauer M.D., Ph.D., MBA, Director of the Institute, Paracelsus Medical University
Other Study IDs: UISM-11
Record Dates: First submitted 2017-10-17; First posted 2018-03-13 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Cardiovascular Diseases
Keywords: outpatient cardiac rehabilitation, exercise training,
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Physical activity — 50min of endurance training combined with 50min of calisthenics; 1-3x/wekk; 6weeks up to 1year

SUMMARY:
Aim of this study is to give evidence to outpatient cardiac rehabilitation in Austria. The database created in this context is supposed to pave the way as instrument to document and comprehend quality of outpatient cardiac rehabilitation in Austria as a key for quality management. Analyses of the created database should be made on a regular basis.

ELIGIBILITY:
Inclusion Criteria:

Any patient who meets inclusion criteria for outpatient cardiac rehabilitation in Austria -

Exclusion Criteria:

* Medical conditions which prevent patients from complying with the exercise program
* Acute infections
* Hypertrophic cardiomyopathy
* Pulmonary artery embolism or phlebothrombosis within the previous 6 months
* Unstable angina pectoris
* Heart failure (NYHA IV)
* Hemodynamically unstable arrhythmia

Ages: 12 Years to 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who qualified for an outpatient cardiac rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Physical Work Capacity (PWC) in Phase II rehabilitation | 6 weeks
  PWC is measured by a graded exercise test on a cycle ergometer at start and end of outpatient cardiac rehabilitation
Change from baseline in Physical Work Capacity (PWC) in Phase III rehabilitation | 1 year
  PWC is measured by a graded exercise test on a cycle ergometer at start and end of outpatient cardiac rehabilitation

SECONDARY OUTCOMES:
Change from baseline in Cholesterol in Phase II rehabilitation | 6 weeks
  Venous blood samples are taken to assess Cholesterol
Change from baseline in Cholesterol in Phase III rehabilitation | 1 year
  Venous blood samples are taken to assess Cholesterol
Change from baseline in Triglycerides in Phase II rehabilitation | 6 weeks
  Venous blood samples are taken to assess Triglycerides
Change from baseline in Triglycerides in Phase III rehabilitation | 1 year
  Venous blood samples are taken to assess Triglycerides
Change from baseline in Blood Glucose in Phase II rehabilitation | 6 weeks
  Venous blood samples are taken to assess blood glucose
Change from baseline in Blood Glucose in Phase III rehabilitation | 1 year
  Venous blood samples are taken to assess blood glucose

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Josef Niebauer, MD, PhD, MBA, Study Chair — Institute of Sports Medicine, Prevention and Rehabilitation Paracelsus Medical University Salzburg, Austria
Locations (1):
- Institute of Sports Medicine, Prevention and Rehabilitation, Paracelsus Medical University, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Niebauer J, Hambrecht R, Velich T, Hauer K, Marburger C, Kalberer B, Weiss C, von Hodenberg E, Schlierf G, Schuler G, Zimmermann R, Kubler W. Attenuated progression of coronary artery disease after 6 years of multifactorial risk intervention: role of physical exercise. Circulation. 1997 Oct 21;96(8):2534-41. doi: 10.1161/01.cir.96.8.2534. PMID 9355890
- [Background] Adams V, Reich B, Uhlemann M, Niebauer J. Molecular effects of exercise training in patients with cardiovascular disease: focus on skeletal muscle, endothelium, and myocardium. Am J Physiol Heart Circ Physiol. 2017 Jul 1;313(1):H72-H88. doi: 10.1152/ajpheart.00470.2016. Epub 2017 May 5. PMID 28476924
- [Result] Niebauer J, Mayr K, Harpf H, Hofmann P, Muller E, Wonisch M, Pokan R, Benzer W. Long-term effects of outpatient cardiac rehabilitation in Austria: a nationwide registry. Wien Klin Wochenschr. 2014 Mar;126(5-6):148-55. doi: 10.1007/s00508-014-0527-3. Epub 2014 Mar 11. PMID 24615677
- See also: Paracelsus Medical University Salzburg, Austria — http://www.pmu.ac.at
- See also: Institute of Sports Medicine, Prevention and Rehabilitation — http://www.salk.at/sportmedizin.html